CLINICAL TRIAL: NCT00711074
Title: An Open-Label, Phase I Study to Assess the Excretion of Radioactivity, Metabolic Profiles and Pharmacokinetics Following a Single Oral Dose of [14C]AZD5672 in Healthy Male Volunteers
Brief Title: Mass Balance and Metabolic Profiling of [14C]AZD5672 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Layton, MD, MRCP(UK), MFPM, Medical Science Director, Early Development RITA, AstraZeneca Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1710C00010; 2008-001528-30 (EUdract No)
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Rheumatoid Arthritis
Keywords: pharmacokinetics; mass balance; radiolabel; AZD5672
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(1-(3-(3,5-difluorophenyl)-3-(4-methanesulfonylphenyl)propyl)piperidin-4-yl)-N-ethyl-2-(4-methanesulfonylphenyl)acetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD5672

INTERVENTIONS:
Drug: AZD5672 — single dose 200mg aqueous solution

SUMMARY:
The purpose of this study is to determine how the body breaks down and excretes the investigational drug, AZD5672.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index (BMI) 18-30 kg/m2, inclusive.
* Clinically normal findings in physical examination, ECG, vital signs, clinical chemistry, haematology & urinalysis, as judged by the investigator

Exclusion Criteria:

* Healthy volunteers who have been exposed to radiation levels above background (eg through X-ray examination) of >5 mSv in the last year, >10 mSv over the last 5 years or a cumulative total of >1 mSv per year of life
* Clinically significant illness within the 2 weeks prior to dosing, as judged by the investigator
* Use of prescribed medication (including St. John's Wort) during the 3 weeks prior to dosing or use of over the counter drugs (including herbals, vitamins and minerals) during 1 week prior to dosing (other than occasional paracetamol use)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2008-06; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
total radioactivity in plasma, whole blood, faeces and urine. | Pre-dose, post dose, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2, 3, 4, 6, 9, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240h
Additional metabolite identification | 0.5h, 3h, 6h, 12h, 24h

SECONDARY OUTCOMES:
general safety assessments: AE reporting, physical examination, ECG, safety haematology and clinical chemistry assessment, vital signs | Screening, pre-dose, Visit 2 (residential period) and visit 3 follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, Study Director — AstraZeneca; Raj Chetty, Principal Investigator — AstraZeneca
Locations (1):
- Research Site, Macclesfield, Cheshire, United Kingdom